CLINICAL TRIAL: NCT03882814
Title: The Effect of Pethidine Analgesia on Labor Duration and Maternal-Fetal Outcomes
Brief Title: Pethidine Analgesia on Labor Duration
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.37
Record Dates: First submitted 2019-03-17; First posted 2019-03-20 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Labor Pain
Keywords: Analgesia; labor; pethidine; Active Phase
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Meperidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pethidine group / study group: Study group; patients given pethidine; The partogram was recorded during delivery. Cervical examination was performed at 2 hour intervals. Recorded in the file. 4 cm and greater cervical dilatation; 50 mg intramuscular (IM) injection was given to pethidine. 200 Montevideo units uterine contractions were reached. Maternal vital signs, maternal complications and neonatal APGAR scores were recorded by the clinician 0-5-15-30-45-60 minutes after pethidine injection.
  Interventions: Drug: pethidine
- control group: The patients who received placebo injection were included in the control group. Saline was given in placebo.
  Interventions: Drug: Placebo - Concentrate

INTERVENTIONS:
Drug: pethidine — Pethidine 50 mg intramuscular (IM) injection was performed when cervical dilatation was at or greater than 4 cm and the cardiotocogram uterine contraction recordings of 200 Montevideo units was reached. Opioid analgesia (pethidine HCl - 50 mg I.M.) was given following amniotomy.
  Groups: Pethidine group / study group
Drug: Placebo - Concentrate — Intramuscular saline was administered to the control group as placebo. Salin intramuscular (IM) injection was performed when cervical dilatation was at or greater than 4 cm and the cardiotocogram uterine contraction recordings of 200 Montevideo units was reached. salon was given following amniotomy.
  Groups: control group

SUMMARY:
Although opioid analgesics are used to treat labor pain, there are still concerns about their side effects.

The researchers in this study; aimed to evaluate the effect of pethidine on active phase duration of labor, labor pain and maternal-neonatal.

50 mg pethidine will be administered intramuscularly to the cases to be included in the study group. The patients in the control group will be given placebo injections.

Vital signs of all cases included in the study will be checked at 0, 5, 15, 30, 45 and 60 minutes. Pain will also be assessed by Visual Analogue Scale (VAS) before injection and at the 1st and 2nd hour after injection. Delivery times, maternal side effects, neonatal apgar scores and fetal findings will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* nullipar-multiparous patients;
* singleton pregnancies 37- 41 weeks (by the last menstrual period).

Exclusion Criteria:

* maternal respiratory rate < 8 /min,
* maternal bradycardia (<60 bpm),
* major fetal congenital anomalies,
* uterine scar presence from previous pregnancies,
* malpresentation,
* antepartum hemorrhage,
* multiple pregnancy,
* labor induction,
* chronic systemic disease,
* rupture fetal membranes,
* epidural analgesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Inclusion criteria were nulliparous and multiparous patients with singleton pregnancies between 37 and 41 completed weeks (according to last menstrual period).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Active phase of labor with pethidine | during labor
  The study group that accepted pethidine injection comprised of 132 patients; The active phase duration was evaluated in minutes.
Labor pain with pethidine | during labor
  Labor pain VAS scores were determined in both groups just prior to pethidine injection (0.hour), and 1st and 2nd hours after injection.
  The VAS scale represents pain with a score of 1 to 10. patients scored points on this scale and these scores were recorded.
  1 point shows the least pain, 10 points the most-irresistible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Kadirogullari P, Yalcin Bahat P, Sahin B, Gonen I, Seckin KD. The Effect of Pethidine Analgesia on Labor Duration and Maternal-Fetal Outcomes. Acta Biomed. 2021 May 12;92(2):e2021065. doi: 10.23750/abm.v92i2.10905. PMID 33988155